CLINICAL TRIAL: NCT06951932
Title: Evaluation of the Impact of Medium-chain Fatty Acids in the Evolution of Newly Diagnosed Mild Cognitive Impairment: Prospective Randomized Controlled Trial
Brief Title: Evaluation of the Impact of Medium-chain Fatty Acids in the Evolution of Newly Diagnosed Mild Cognitive Impairment
Acronym: MCI-MCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASO.MedI.23.02
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Montreal Cognitive Assessment; medium-chain triglycerides
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a nonpharmacological dietary supplement interventional study, controlled, randomized with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean-type food regimen using extra virgin olive oil (Active Comparator): Patients with with first diagnosis of MCI referred to the S.C of Neurology and/or Geriatrics and/or Internal Medicine of the SS. Antonio e Biagio e Cesare Arrigo of Alessandria University Hospital, randomized into the control arm
  Interventions: Other: Mediterranean-type food regimen using extra virgin olive oil
- Mediterranean-type diet with MCT supplementation (Experimental): Patients with with first diagnosis of MCI referred to the S.C of Neurology and/or Geriatrics and/or Internal Medicine of the SS. Antonio e Biagio e Cesare Arrigo of Alessandria University Hospital, randomized into the experimental arm
  Interventions: Dietary Supplement: Mediterranean-type diet with MCT supplementation

INTERVENTIONS:
Dietary Supplement: Mediterranean-type diet with MCT supplementation — The treatment arm will follow a Mediterranean diet supplemented by daily intake of MCT (30 mL)
  Arms: Mediterranean-type diet with MCT supplementation
Other: Mediterranean-type food regimen using extra virgin olive oil — The arm will follow a Mediterranean diet with an indication to take extra virgin olive oil as the main fat in the diet daily
  Arms: Mediterranean-type food regimen using extra virgin olive oil

SUMMARY:
Mild cognitive impairment (MCI) is considered the intermediate stage between the changes observed in physiological aging and dementia. Currently, there is no drug therapy, and available drugs offer only minimal benefit on symptoms, only partially slowing the course of the condition. Studies in the literature have investigated the role of omega-3 fatty acids in MCI, and when administered over a period of six months, they appear to improve clinical condition and mood. In addition, medium-chain triglycerides (MCTs) appear to exert an antioxidant function, enhance cognitive ability in patients with MCI or Alzheimer's, and promote deep sleep state.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is considered the intermediate stage between the changes observed in physiological aging and dementia. The need to diagnose MCI at an early stage is driven by the hypothesis that therapeutic interventions may be more effective in the early stages of the disease. In addition, many studies have shown that sleep disturbances can affect neurodegeneration and be used as a marker of disease, manifesting before cognitive impairment itself. Currently, there is no drug therapy, and available drugs offer only minimal benefit on symptoms, only partially slowing the course of the condition. Studies in the literature have investigated the role of omega-3 fatty acids in MCI, and when administered over a period of six months, they appear to improve clinical condition and mood. In addition, medium-chain triglycerides (MCTs) appear to exert an antioxidant function, enhance cognitive ability in patients with MCI or Alzheimer's, and promote deep sleep state

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years;
* Diagnosis of MCI;
* Disease duration of less than 24 months from symptom onset;
* Absence of malnutrition (diagnosed according to the NRS 2002 screening test) and with oral intakes sufficient to cover energy requirements (calculated by the Harris-Benedict formula, adjusted for activity factor and pathology);
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Patients on total or supplemental enteral nutrition
* Severe dysphagia
* Patients with glycated hemoglobin > 8%
* Patients on insulin therapy
* Patients with poor beta-cell function (e.g., pancreasectomy, acute and chronic pancreatitis)
* Patients with liver failure: MELD score > 9
* Malnutrition (diagnosed according to the NRS 2002 screening test) and with per os intakes < 60% of energy requirements (calculated using the Harris-Benedict formula, corrected for activity factor and pathology)
* Metabolic disorders and/or enzyme disorders, dyslipidemia with total cholesterolemia >300 mg/dl and/or triglyceridemia >400 mg/dl)
* Acute inflammatory disease or ongoing or recent (within 30 days) infectious states
* Hypo- and hyperthyroidism not adequately compensated by treatment
* Heart failure (NYHA III-IV), unstable angina, recent (<6 months) acute cardiovascular or cerebrovascular events
* Pregnancy or lactation
* Neurological disorders other than MCI, psychiatric disorders
* Nutrition and eating disorder
* Alcohol abuse
* Institutionalized patients
* Participation in experimental therapies in the 2 months prior to enrollment
* Allergy to MCT oil, nuts

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Effect of medium-chain triglycerides (MCT) intake on cognitive impairment | 6 months after baseline
  Evaluate the effect of medium-chain triglycerides (MCT) intake on cognitive decline in patients with first diagnosis of MCI through the use of the Montreal Cognitive Assessment (MoCA), that includes a series of tests of visuospatial/executive functions, naming, attention, language, abstraction, delayed recall, and orientation for a total score of 30 (best cognitive status).

SECONDARY OUTCOMES:
Positive effect of MCT intake on sleep quality | Baseline and 6 months after baseline
  Evaluate the positive effect of MCT intake on sleep quality in patients with MCI using the Pittsburgh and Epworth Scales, sleep quality rating scales.
Evaluation of quality of life | Baseline, 3 months after baseline and 6 months after baseline
  Assessing quality of life through the QoL AD score (Quality of life in Alzheimer's Disease), characterized by 15 items that can be answered by choosing from four options that are scored from 1 (poor) to 4 (excellent). The total score ranges from 13 (worst quality of life) to 52 (best quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No